CLINICAL TRIAL: NCT05515354
Title: Coordinating Smoking Cessation Treatment With Menstrual Cycle Phase to Improve Quit Outcomes: A Randomized Controlled Trial
Brief Title: Smoking Cessation and Menstrual Cycle Phase
Acronym: MC-NRT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Cancer Society (CCS) (Other)
Responsible Party: Principal Investigator, Laurie Zawertailo, Senior Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 022-2022
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Nicotine Dependence; Tobacco Smoking; Smoking Cessation; Nicotine Use Disorder; Substance Use Disorders
Keywords: Menstrual Cycle; Ovarian Hormones; Smoking Cessation Treatment; Nicotine Replacement Therapy; Cancer Prevention; Randomized Controlled Trial; Estrogen; Progesterone
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Smoking; Smoking Cessation; Substance-Related Disorders | interventions — Nicotine Replacement Therapy; Tobacco Use Cessation Devices; Nicotine Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mid-Follicular Phase Target Quit Date (Experimental): Participants will start their quit attempts during the mid-follicular phase of their MC (6-8 days post-onset of menses). Each participant will be provided with a range of appropriate dates based on the information about their menstrual cycle, and they will select a target quit date from the range. Participants will be receiving NRT and will have access to behavioral support for the following 6 weeks.
  Interventions: Other: Timing of nicotine replacement therapy start date; Drug: Nicotine Replacement Therapy Agent
- Mid-Luteal Phase Target Quit Date (Experimental): Participants will start their quit attempts during the mid-luteal phase of their MC (6-8 days pre-onset of menses). Each participant will be provided with a range of appropriate dates based on the information about their menstrual cycle, and they will select a target quit date from the range. Participants will be receiving NRT and will have access to behavioral support for the following 6 weeks.
  Interventions: Other: Timing of nicotine replacement therapy start date; Drug: Nicotine Replacement Therapy Agent
- Randomly Selected Target Quit Date (Usual Care) (Active Comparator): Participants will start their quit attempts within 30 days of their enrollment into the study. They will select their target quit dates without regard for their MC. Participants will be receiving NRT and will have access to behavioral support for the following 6 weeks.
  Interventions: Drug: Nicotine Replacement Therapy Agent

INTERVENTIONS:
Other: Timing of nicotine replacement therapy start date — Nicotine replacement therapy and abstinence from smoking are initiated at a specific period with regard to the menstrual cycle.
  Other Names: Timing of target quit date
  Arms: Mid-Follicular Phase Target Quit Date; Mid-Luteal Phase Target Quit Date
Drug: Nicotine Replacement Therapy Agent — Nicotine patch and a choice of nicotine gum or lozenge (2 mg) for 6 weeks. Participants who smoke 10 or more cigarettes per day receive a package of 21 mg, 14 mg, and 7 mg nicotine patches. For participants who smoke 5-9 (inclusive) cigarettes per day, the package contains 14 mg and 7 mg nicotine patches.
  Other Names: Nicotine Patch; Nicotine Gum; Nicotine Lozenge

SUMMARY:
Tobacco use is a risk factor for at least 20 types of cancer and remains the leading preventable cause of cancer in Canada. Smoking cessation is an important cancer prevention strategy for the close to 2 million Canadian women who currently smoke. However, findings from controlled trials and real-world clinical settings indicate that women have greater difficulty achieving abstinence following a quit attempt than men. There is some evidence that hormonal levels and fluctuations throughout the menstrual cycle (MC) may contribute to the greater difficulty women experience when trying to quit smoking. In this study, the start of a quit attempt using nicotine replacement therapy (NRT) will be targeted to specific phases of MC. It was hypothesized that starting a quit attempt during the first half of MC (follicular phase) will result in increased quit success compared to starting during the second half of MC (luteal phase) or the usual practice of not targeting quit start date to MC phase.

DETAILED DESCRIPTION:
Evidence for the influence of the menstrual cycle (MC) phase on smoking cessation outcomes is contradictory and has been limited by small samples and a lack of clarity surrounding ideal quit date timing. Therefore, this large rigorously designed study aims to clarify whether targeting quit date to either the follicular or luteal phase of MC improves quit success. The primary hypothesis states that participants assigned a TQD in the follicular phase of their MC will be more likely to have quit successfully on day 7 of treatment than participants setting their own TQD (usual care). Quit rates at the end of treatment and 6 months post-TQD were identified as secondary objectives.

Participants will enroll in an online smoking cessation program providing nicotine replacement therapy (NRT) and behavioral support. Participants will receive a 6-week supply of NRT consisting of nicotine patch plus their choice of nicotine gum or lozenge, which the participants will be instructed to start on their target quit date (TQD). Eligible individuals will be randomized to a TQD: [1] during the mid-luteal phase of their MC (6-8 days pre-onset of menses), [2] during the mid-follicular phase of their MC (6-8 days post-onset of menses), or [3] within 30 days of enrollment with no regard to MC phase (usual care). Behavioural support will consist of a free downloadable app (My Change Plan) and brief videos delivered via e-mail. These videos will be produced by the CAMH Nicotine Dependence Service and will focus on health behavior change strategies such as building a quit plan, coping with cravings, and relapse prevention.

ELIGIBILITY:
Inclusion Criteria:

* Must provide informed consent following the CAMH REDCap e-consent framework and procedures;
* Stated willingness to comply with all study procedures;
* Naturally cycling individuals with regular MCs (defined as length ranging 21 to 35 days over past 6 months);
* Daily smoker of ≥5 cigarettes per day (CPD) over past 6 months;
* Intention to quit smoking within the next 30 days and willing to make a quit attempt on their assigned TQD;
* Interested in using, and able to use, nicotine patches and gum or lozenge as a smoking cessation aid;
* Willing to provide a valid e-mail address to be used for study communications and to complete online questionnaires.

Exclusion Criteria:

* Current use of progesterone, estrogen, testosterone, or fertility treatment;
* Current use of nicotine replacement therapy or other smoking cessation medications (e.g., varenicline, bupropion);
* Use of hormonal contraceptives in the past 6 months (e.g., pill, patch, hormonal intrauterine device [IUD], ring);
* Pregnancy, or trying to become pregnant in the next 2-3 months;
* Known hypersensitivity or allergies to any of the components of the nicotine patch;
* Daily or almost daily use of cannabis in the past 6 months;
* Daily or almost daily use of tobacco or nicotine products other than cigarettes (e.g., smokeless tobacco, heat-not-burn products, e-cigarettes) in the past 6 months;
* Polycystic ovary syndrome diagnosis;
* Unstable psychiatric condition (including substance use disorder) which would compromise study compliance;
* Life threatening arrhythmias or severe/worsening angina pectoris;
* Myocardial infarction or cerebral vascular accident in the past 2 weeks; or
* Diagnosed with a terminal illness.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1200 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
7-day point prevalence of abstinence | 7 days post-target quit date
  Proportion of the sample that has been abstinent from smoking for 7 days at the time of assessment (i.e., managed to quit smoking on their target quit date).

SECONDARY OUTCOMES:
End-of-treatment 7-day point prevalence of abstinence | 6 weeks post-target quit date
  Proportion of the sample that has been abstinent from smoking for at least 7 days at the time of assessment.
Follow-up 7-day point prevalence of abstinence | 6 months post-target quit date
  Proportion of the sample that has been abstinent from smoking for at least 7 days at the time of assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie A Zawertailo, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Nicotine Dependence Clinic, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Carpenter MJ, Saladin ME, Leinbach AS, Larowe SD, Upadhyaya HP. Menstrual phase effects on smoking cessation: a pilot feasibility study. J Womens Health (Larchmt). 2008 Mar;17(2):293-301. doi: 10.1089/jwh.2007.0415. PMID 18321181
- [Background] Franklin TR, Ehrman R, Lynch KG, Harper D, Sciortino N, O'Brien CP, Childress AR. Menstrual cycle phase at quit date predicts smoking status in an NRT treatment trial: a retrospective analysis. J Womens Health (Larchmt). 2008 Mar;17(2):287-92. doi: 10.1089/jwh.2007.0423. PMID 18321180
- [Background] Piper ME, Cook JW, Schlam TR, Jorenby DE, Smith SS, Bolt DM, Loh WY. Gender, race, and education differences in abstinence rates among participants in two randomized smoking cessation trials. Nicotine Tob Res. 2010 Jun;12(6):647-57. doi: 10.1093/ntr/ntq067. Epub 2010 May 3. PMID 20439385
- [Background] Poirier AE, Ruan Y, Grevers X, Walter SD, Villeneuve PJ, Friedenreich CM, Brenner DR; ComPARe Study Team. Estimates of the current and future burden of cancer attributable to active and passive tobacco smoking in Canada. Prev Med. 2019 May;122:9-19. doi: 10.1016/j.ypmed.2019.03.015. PMID 31078177
- [Background] Saladin ME, McClure EA, Baker NL, Carpenter MJ, Ramakrishnan V, Hartwell KJ, Gray KM. Increasing progesterone levels are associated with smoking abstinence among free-cycling women smokers who receive brief pharmacotherapy. Nicotine Tob Res. 2015 Apr;17(4):398-406. doi: 10.1093/ntr/ntu262. PMID 25762749
- [Background] Smith PH, Bessette AJ, Weinberger AH, Sheffer CE, McKee SA. Sex/gender differences in smoking cessation: A review. Prev Med. 2016 Nov;92:135-140. doi: 10.1016/j.ypmed.2016.07.013. Epub 2016 Jul 26. PMID 27471021
- [Background] Statistics Canada. (2020). Smokers, by age group. Retrieved August 23, 2021, from https://www150.statcan.gc.ca/t1/tbl1/en/tv.action?pid=1310009610&pickMembers%5B0%5D=1.1&pickMembers%5B1%5D=3.3&cubeTimeFrame.startYear=2018&cubeTimeFrame.endYear=2019&referencePeriods=20180101%2C20190101
- [Background] World Health Organization. (2020). Who report on cancer: Setting priorities, investing wisely and providing care for all. World Health Organization. Retrieved August 12, 2022, from https://www.who.int/publications-detail-redirect/9789240001299
- [Background] Weinberger AH, Smith PH, Allen SS, Cosgrove KP, Saladin ME, Gray KM, Mazure CM, Wetherington CL, McKee SA. Systematic and meta-analytic review of research examining the impact of menstrual cycle phase and ovarian hormones on smoking and cessation. Nicotine Tob Res. 2015 Apr;17(4):407-21. doi: 10.1093/ntr/ntu249. PMID 25762750
- [Derived] Zawertailo L, Kabir T, Voci S, Tanzini E, Attwells S, Malat L, Veldhuizen S, Minian N, Dragonetti R, Melamed OC, Mei-Dan E, Selby P. Coordinating smoking cessation treatment with menstrual cycle phase to improve quit outcomes (MC-NRT): study protocol for a randomized controlled trial. Trials. 2023 Apr 1;24(1):251. doi: 10.1186/s13063-023-07196-1. PMID 37005655